CLINICAL TRIAL: NCT07238842
Title: A Non-inferiority Study of the Virtual Agent-based Versus Teacher-led Psychological Literacy Enhancement Method in Improving Adolescents' Mental Health Literacy
Brief Title: Non-inferiority of Virtual vs. Traditional Methods in Adolescent Mental Health Literacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MZhao-024
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teacher-Led Psychological Literacy Instruction (Active Comparator): Participants in this arm receive the identical 6-week psychological literacy curriculum, but delivered by trained school psychology teachers through traditional face-to-face classroom instruction. Each weekly session lasts 45-60 minutes and follows the same structure and content as the virtual agent arm, including the same four thematic modules. Teachers use standard pedagogical methods such as lectures, group discussions, role-playing, and worksheet activities. This arm serves as the active control condition, representing the current standard of school-based mental health education in China.
  Interventions: Behavioral: Teacher-Led Psychological Literacy Instruction
- Virtual Agent-Delivered Psychological Literacy Program (Experimental): Participants in this arm receive a 6-week psychological literacy curriculum delivered entirely by an AI-powered virtual digital agent. The program consists of weekly 45-60 minute interactive sessions aligned with China's national guidelines for mental health education (e.g., Guidelines for Mental Health Education in Primary and Secondary Schools, 2012). The content covers four core modules: (1) psychological foundations and self-awareness, (2) stress and challenge coping skills, (3) interpersonal and communication skills, and (4) healthy lifestyle and future planning. The virtual agent uses scripted but adaptive dialogue, emotion-aware responses, and multimedia engagement to deliver the same evidence-based curriculum used in the control arm. Sessions are conducted in a classroom setting using school-provided computers.
  Interventions: Behavioral: Virtual Agent-Delivered Psychological Literacy Training

INTERVENTIONS:
Behavioral: Teacher-Led Psychological Literacy Instruction — This intervention delivers the identical 6-week psychological literacy curriculum as the virtual agent arm, but through standard face-to-face instruction by certified school psychology teachers. Teachers follow a detailed manualized lesson plan covering the same four thematic modules and learning objectives. Sessions include traditional pedagogical techniques such as didactic teaching, group discussion, role-playing exercises, reflective writing, and in-class activities. Each session lasts 45-60 minutes and occurs weekly in the regular classroom setting. Teachers are trained to adhere to the protocol to ensure content equivalence with the virtual agent condition, though minor natural variations in delivery style, pacing, or classroom interaction may occur. This intervention represents the current standard of practice for school-based mental health education in China and serves as the active control condition.
  Arms: Teacher-Led Psychological Literacy Instruction
Behavioral: Virtual Agent-Delivered Psychological Literacy Training — This intervention consists of a 6-week, school-based psychological literacy program delivered by an AI-powered virtual digital agent. The agent uses real-time animation, speech synthesis, and scripted but context-sensitive dialogue to guide students through evidence-based mental health content aligned with China's national mental health education guidelines. The curriculum includes four modules: (1) psychological foundations and self-awareness, (2) stress and coping skills, (3) interpersonal and family communication, and (4) healthy digital habits, sleep, and future planning. Each weekly session (45-60 minutes) is fully digital, interactive, and delivered via classroom computers. The virtual agent maintains consistent content fidelity across all participants. This intervention leverages AI technologies-including natural language understanding and emotion-aware feedback-but does not provide clinical therapy or real-time personalized adaptation beyond pre-programmed branching logic.
  Arms: Virtual Agent-Delivered Psychological Literacy Program

SUMMARY:
The goal of this clinical trial is to determine whether a digital psychological literacy program delivered by an AI-powered virtual agent is non-inferior to traditional teacher-led instruction in improving mental health literacy among adolescents. The study focuses on middle and high school students aged 11 to 18 years attending a school in Shanghai, China, including those with varying levels of emotional well-being but excluding those with diagnosed psychiatric disorders or severe physical illness.

The main questions it aims to answer are:

Is the virtual agent-delivered psychological literacy program as effective as teacher-led instruction in improving adolescents' mental health literacy? Does the virtual agent intervention lead to comparable or better outcomes in secondary measures such as depression, anxiety, psychological resilience, sleep quality, and digital well-being?

Researchers will compare students receiving 6 weekly sessions from a virtual digital agent to students receiving the same curriculum delivered by trained psychology teachers to see if the AI-based approach achieves similar improvements in mental health knowledge, attitudes, and help-seeking behaviors.

Participants will:

Complete online assessments at baseline, week 3, week 6 and week 18 covering mental health literacy (UMHL-A), depression (PHQ-9), anxiety (GAD-7), psychological resilience (RSCA), and other well-being indicators Attend one 45-60 minute session per week for 6 weeks, either interacting with the virtual agent or participating in a teacher-led class Optionally take part in a brief satisfaction survey and/or a focus group interview after the intervention to share their experiences

ELIGIBILITY:
Inclusion Criteria:

1. Age between 11 and 18 years inclusive.
2. Able to fluently operate a computer or smartphone.
3. Possess normal language expression and reading comprehension abilities.
4. Voluntarily agree to participate in the study and provide signed informed consent (and parental consent where required by local regulations).

Exclusion Criteria:

1. Diagnosed with a psychiatric disorder that impairs the ability to complete assessments or participate in the intervention.
2. Suffering from a severe physical illness, central nervous system disease, or substance use disorder that could interfere with study participation or outcomes.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Adolescent Mental Health Literacy | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Mental health literacy is assessed using the UMHL-A (Adolescent Mental Health Literacy Scale), a validated Chinese-language instrument that evaluates two key domains:
  Part A: Knowledge and understanding of mental health concepts, common psychological problems, risk/protective factors, and help-seeking resources.
  Part B: Attitudes toward mental health issues and behavioral intentions to seek help or support others.
  Higher total scores indicate greater mental health literacy. The scale has demonstrated strong reliability and validity in Chinese adolescent populations.

SECONDARY OUTCOMES:
Change in Depressive Symptom Severity | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Depressive symptoms are measured using the PHQ-9 (Patient Health Questionnaire-9), a widely used 9-item self-report scale that assesses the frequency of core depression symptoms (e.g., low mood, anhedonia, sleep disturbance) over the past two weeks. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), yielding a total score from 0 to 27. Higher scores indicate more severe depressive symptoms. The Chinese version has established reliability and clinical utility.
Change in Anxiety Symptom Severity | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Anxiety symptoms are assessed using the GAD-7 (Generalized Anxiety Disorder-7), a 7-item self-report questionnaire that measures the frequency of anxiety symptoms (e.g., excessive worry, restlessness, difficulty controlling worry) over the past two weeks. Scores range from 0 to 21, with higher scores indicating greater anxiety severity. The Chinese version is well-validated for use in adolescents.
Change in Psychological Resilience | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Psychological resilience is evaluated using the RSCA (Resilience Scale for Chinese Adolescents), a culturally adapted scale that measures adolescents' capacity to adapt positively in the face of adversity. It assesses domains such as self-efficacy, emotional regulation, goal orientation, and perceived social support. Higher scores reflect greater resilience.
Change in Behavioral and Emotional Difficulties | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Emotional and behavioral problems are screened using the SDQ (Strengths and Difficulties Questionnaire), specifically the subscales for emotional symptoms, conduct problems, hyperactivity, peer relationship issues, and prosocial behavior. The total difficulties score (range: 0-40) is used as a global indicator of psychosocial adjustment. The Chinese adolescent version is reliable and commonly used in school settings.
Change in Sleep Quality | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Sleep quality over the past month is assessed using the PSQI (Pittsburgh Sleep Quality Index), a 19-item self-report instrument that evaluates seven dimensions: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Total scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Change in Risk of Gaming Disorder | From baseline to the end of the 6-week intervention period, and at 3-month follow-up
  Risk of gaming disorder is measured using the GDSS (Gaming Disorder Screening Scale), an 18-item Likert-type scale based on DSM-5 and ICD-11 criteria. It assesses symptoms such as loss of control over gaming, prioritizing gaming over other activities, and continued use despite negative consequences. Total scores range from 18 to 72, with higher scores indicating greater risk.
Change in Adolescent Mental Health Literacy at 3-Month Follow-Up | From baseline to 3 months after the end of the 6-week intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Nanhui No.2 Middle School, Shanghai, China